CLINICAL TRIAL: NCT04352374
Title: Effect of Aerobic Exercises Versus Device Guided Breathing on Gestational Hypertension
Brief Title: Aerobic Exercises vs Device Guided Breathing on Gestational Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Aly Elbandrawy, Prof faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cairo university P.T
Record Dates: First submitted 2020-04-12; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Hypertension ,Pregnancy
Keywords: Hypertension; Pregnancy; Aerobic exercise; Device guided breathing
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A total of 75 participants were initially screened. After the screening process, 60 participants were found to be eligible to participate in the study. In total, 50 (100%) participants completed the treatment program
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pregnant women were randomized using an opaque sealed envelope that was sequentially numbered and statistically generated by a computer program. The envelope contained information about the random allocation group: group (A), engaged in aerobic exercise twice a week under the supervision of a physical therapist, and group (B), engaged in device guided breathing exercises. Both groups received antihypertensive medications. Random allocation of the subjects was performed by another investigator, who did not participate directly in the research study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Experimental): The therapist advised all participants of this group to drink a plenty of water before and after the exercise session to avoid excessive loss of body water during the session. Pregnant women were instructed to have a light meal about one hour before the performance of exercise and to wear comfortable clothes.
  Participants in this group were given a Low-Intensity Aerobic Exercise with Borg scale RPE at 11. Participants were asked to maintain this intensity of rate of perceived exertion throughout the 45 minutes' duration of the aerobic training.
  During the training session, the therapist stood near the patient to observe and detect signs of stopping the exercise. The therapist continuously asked the patient if she felt pain, dizzy or shortens of breath.
  No complications were observed during physical exercise sessions, for example, hypertensive crisis, hypotension, hyperthermia, musculoskeletal lesions, or other complications identified that demanded interruption of the exercise.
  Interventions: Other: Aerobic exercise
- Device guided breathing group (Active Comparator): At the beginning the researcher explained the device and study procedures to every participant of this group .The device consists of a control box, headphones and a respiratory rate monitor attached as a sensor belt around the user's chest.
  The participant is instructed to alter their breathing rate, aiming for up to 10 breaths per minute, in response to a melody played to them via the asked to use the device for at least 40 min per week, with each session lasting at least 10 min
  Interventions: Device: Device guided breathing

INTERVENTIONS:
Other: Aerobic exercise — a Low-Intensity Aerobic Exercise with Borg scale RPE at 11.
  Arms: Aerobic exercise group
Device: Device guided breathing — The device consists of a control box, headphones and a respiratory rate monitor attached as a sensor belt around the user's chest.
  Arms: Device guided breathing group

SUMMARY:
Aim To compare between the effect of aerobic exercise versus device guided breathing (DGB) on blood pressure in gestational hypertensive patients. Participants and Methods Randomized controlled trial, which included 60 singleton pregnant women (at 21-week gestation) diagnosed with gestational hypertension. They were divided into two groups: group (A) received aerobic exercise with a treadmill twice a week, for 45 minutes; and group (B) received Device guided breathing exercise for at least 40 min per week, with each session lasting at least 10 min. Assessment of the systolic blood pressure (SBP) and diastolic blood pressure (DBP) for all participants in the two studied groups (A, B) was carried out at begining of the study and at week-36 of gestation with mercury column sphygmomanometer.

DETAILED DESCRIPTION:
Sixty singleton pregnant women, diagnosed with gestational hypertension (GH) at 21- week of gestation, and aged between 25-35 years were randomized. GH was defined as blood pressure higher than 140/90 measured on two separate occasions, more than 6 hours apart, without the presence of protein in the urine and diagnosed after 20 weeks of gestation.

Women with multiple pregnancies, cervical insufficiency, vaginal bleeding, heart disease, systemic lupus erythematosus, kidney failure, and neurologic disorders were excluded from the study. For inclusion in the study, pregnant women also could not be engaged in any supervised physical exercise, at the time of selection and when signing a free written informed consent term.

Pregnant women were randomized using an opaque sealed envelope that was sequentially numbered and statistically generated by a computer program. The envelope contained information about the random allocation group: group (A), engaged in aerobic exercise twice a week under the supervision of a physical therapist, and group (B), engaged in device guided breathing exercises. Both groups received antihypertensive medications. Random allocation of the subjects was performed by another investigator, who did not participate directly in the research study.

Exercise program for group (A) The therapist advised all participants to drink a plenty of water before and after the exercise session to avoid excessive loss of body water during the session. Pregnant women were instructed to have a light meal about one hour before the performance of exercise and to wear comfortable clothes.

Participants in this group were given a Low-Intensity Aerobic Exercise with Borg scale RPE at 11. Participants were asked to maintain this intensity of rate of perceived exertion throughout the 45 minutes' duration of the aerobic training.

During the training session, the therapist stood near the patient to observe and detect signs of stopping the exercise. The therapist continuously asked the patient if she felt pain, dizzy or shortens of breath.

Device guided breathing for group (B) The FDA approved the Resperate device as an adjunct anti-hypertensive treatment approach that guides home users to alter their breathing rate in response to instructed signals .

At the beginning the researcher explained the device and study procedures to every participant of group (B).The device consists of a control box, headphones and a respiratory rate monitor attached as a sensor belt around the user's chest.

The participant is instructed to alter their breathing rate, aiming for up to 10 breaths per minute, in response to a melody played to them via the asked to use the device for at least 40 min per week, with each session lasting at least 10 min .

All pregnant females of both groups were requested to maintain routine lifestyle habits with regard to diet intake throughout the study. All blood pressure measurements were conducted during the morning hours. Arterial blood pressure was measured using a standard mercury sphygmomanometer with appropriate cuff size, after subjects had rested in the sitting position for at least 5 minutes. BP was measured and presented at 20 week gestation and week-36 of gestation. Two readings were taken at 2 minutes interval, and the average values were used as the baseline value.

ELIGIBILITY:
Inclusion Criteria:

* Sixty singleton pregnant women, diagnosed with gestational hypertension (GH) at 21- week of gestation, and aged between 25-35 years were randomized. GH was defined as blood pressure higher than 140/90 measured on two separate occasions, more than 6 hours apart, without the presence of protein in the urine and diagnosed after 20 weeks of gestation.

Exclusion Criteria:

* Women with multiple pregnancies, cervical insufficiency, vaginal bleeding, heart disease, systemic lupus erythematosus, kidney failure, and neurologic disorders were excluded from the study. For inclusion in the study, pregnant women also could not be engaged in any supervised physical exercise, at the time of selection and when signing a free written informed consent term.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gestational hypertension
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Arterial blood pressure | from enrollment to end of treatment at 36 week gestation
  Change in Arterial blood pressure was measured using a standard mercury

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa M Elbandrawy, Assis prof, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No
journal publication, Google Scholar, ResearchGate, LinkedIn